CLINICAL TRIAL: NCT00029315
Title: Intraventricular Rt-PA Pharmacokinetic and Pharmacodynamic Study
Brief Title: Intraventricular Rt-PA in Patients With Intraventricular Hemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FD-R-2018-01; FD-R-002018-01
Record Dates: First submitted 2002-01-10; First posted 2002-01-11 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-12

CONDITIONS: Cerebral Hemorrhage
Keywords: Intraventricular hemorrhage; Subarachnoid hemorrhage; Intracerebral hemorrhage; Pharmacokinetics; Recombinant Proteins; Anticoagulants; Tissue Plasminogen Activator; Pharmacology; Catheters, Indwelling; Cerebral Ventricles
MeSH Terms: conditions — Cerebral Hemorrhage; Subarachnoid Hemorrhage | interventions — Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Recombinant Tissue Plasminogen Activator (rt-PA)

SUMMARY:
This is a study to evaluate how recombinant tissue plasminogen activator (rt-PA) is utilized in patients with intraventricular hemorrhage (IVH). rt-PA is a drug that has been shown to dissolve blood, and may allow intraventricular catheters to be more effective for a longer period of time.

DETAILED DESCRIPTION:
IVH occurs in about 40 percent of intracerebral hemorrhage cases and 15 percent of aneurysmal subarachnoid hemorrhage cases. Evidence supports a strong contribution of IVH to morbidity and mortality after cerebral hemorrhage. External ventricular drainage (EVD) is required clinical management; however, EVD via intraventricular catheter alone fails to prevent much of the morbidity and mortality of IVH. This study seeks to demonstrate the safety and efficacy of intraventricular thrombolysis, using rt-PA, as a method of removing this blood and altering morbidity and mortality. Patients will receive intraventricular injections of rt-PA or placebo every 12 hours. They will be followed prospectively with daily head CT scans during the acute-treatment phase and again between Days 28 and 32.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Intraventricular hemorrhage (IVH) confirmed by CT scan
* More than 12 hours post bleed
* Hematoma size stable by CT scan
* Post-IVH catheter CT scan
* Able to begin study within 24 hours of bleed

Exclusion criteria:

* Infratentorial bleed
* Supratentorial bleed greater than 30 cc
* Unclipped aneurysm suspected
* Arteriovenous malformation suspected
* Any severe, complicating illness (e.g., AIDS or DNR)
* Cardiovascular parameters that could confound study (e.g., myocardial infarction, pulmonary emboli, systemic fibrinolysis)
* Active internal bleeding
* Requirement for heparin doses greater than 10,000 U/day
* Concurrent coumadin
* Known allergy to rt-PA
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-09; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States